CLINICAL TRIAL: NCT04162392
Title: Physical Activity Barriers in Acute Exacerbated COPD
Brief Title: Physical Activity Barriers in AECOPD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Granada (Other)
Responsible Party: Principal Investigator, Marie Carmen Valenza, Principal investigator, Universidad de Granada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DF0084UG
Record Dates: First submitted 2019-11-11; First posted 2019-11-14 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: COPD Exacerbation
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental)
  Interventions: Other: shared decision making
- Control group (Active Comparator)
  Interventions: Other: control group

INTERVENTIONS:
Other: shared decision making — Patients can choose the intervention that they want. There are different physiotherapy interventions were the patients have to do physical activity during the hospital stay. The physiotherapist explains the advantages and disadvantages of each treatment before they choose.
  Arms: Experimental group
Other: control group — Patients receive a physiotherapy intervention but they do not have the opportunity to choose the treatment
  Arms: Control group

SUMMARY:
Chronic obstructive pulmonary disease (COPD) is a leading cause of morbidity and mortality worldwide. Patients require good communication with the physician to improve control illness. Shared decision making is a good option to improve physical activity barriers in acute exacerbated COPD patients during the hospitalization period.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were COPD patients hospitalized due to acute exacerbation

Exclusion Criteria:

* Exclusion criteria were the inability to provide informed consent, the presence of psychiatric or cognitive disorders, progressive neurological disorders, organ failure, cancer, or inability to cooperate. Patients who had experienced another exacerbation of COPD in the previous month were also excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Health related quality of life: EQ-5D | Participants will be followed for the duration of hospital stay, an expected average of 9 days and after discharge 3 months follow up
  European Quality of Life questionnaire consists of the EQ-5D visual analog scale and the EQ-5D index. The visual analog scale has a rating scale of 0-100 (0 worst possible health, and 100 best possible health). The questionnaire has 5 domains: mobility, self-care, usual activity, pain, and anxiety-depression. For each item, the subject selects one of 3 descriptive health states (from good to poor).
Functional capacity | Participants will be followed for the duration of hospital stay, an expected average of 9 days and after discharge 3 months follow up
  The International Physical Activity Questionnaire (IPAQ) short form measures walking, moderate- and vigorous intensity, and total PA and daily time spent sitting on weekdays. PA was reported in MET·minutes/week and days per week and was scored using standardized IPAQ scoring protocols to yield total metabolic equivalent minutes (MET·minutes/week) of PA per week. Sitting time was reported as the amount of time in hours and/or minutes participants spent sitting on a weekday during the past seven days.
Barriers to Being Active Quiz | Participants will be followed for the duration of hospital stay, an expected average of 9 days and after discharge 3 months follow up
  The Barriers to Being Active Quiz is a 21-item scale that provides a measure of 7 self-reported barriers to being physically active.This instrument uses a 4-point Likert scale for individuals to identify if they would say or think any of the statements would be true for them, with 0 being very unlikely to 3 being very likely. Per instrument instructions, each barrier has 3 items that are summed for scoring, with a range of 0 to 9 for each.

IPD SHARING:
Plan to Share IPD: Undecided